CLINICAL TRIAL: NCT01212068
Title: Connectivity Analysis for Investigation of Auditory Impairment in Epilepsy
Status: Terminated | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100211; 10-DC-0211
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-04-04

CONDITIONS: Brain Mapping; Intracranial Central Nervous System Disorder; Epilepsy; Auditory Perceptual Disorder; Hearing Disorder
Keywords: MEG; Epilepsy; Brain Imaging; Brain Scan; Auditory Processing; Auditory Perceptual Disorder
MeSH Terms: conditions — Epilepsy; Auditory Perceptual Disorders; Hearing Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Background:

* People with epilepsy often have auditory processing disorders that affect their ability to hear clearly and may cause problems with understanding speech and other kinds of verbal communication. Researchers are interested in developing better ways of studying what parts of the brain are affected by hearing disorders and epilepsy, and they need better clinical tests to measure how individuals process sound. These tests will allow researchers to examine and evaluate the effects of epilepsy and related disorders on speech and communication.
* A procedure called a magnetoencephalography (MEG) can be used to measure the electrical currents involved in brain activity. Researchers are interested in learning whether MEG can be used to detect differences in the processing of simple sounds in patients with epilepsy, both with and without hearing impairments.

Objectives:

- To measure brain activity in hearing impaired persons with epilepsy and compare the results with those from people with normal hearing and epilepsy as well as people with normal hearing and no epilepsy. This research is performed in collaboration with Johns Hopkins Hospital and epilepsy patients must be candidates for surgery at Johns Hopkins.

Eligibility:

* Individuals between 18 to 55 years of age who (1) have epilepsy and have hearing impairments, (2) have epilepsy but do not have hearing impairments, or (3) are healthy volunteers who have neither epilepsy nor hearing impairments.
* Participants with epilepsy must have developed seizures after 10 years of age, and must be candidates for grid implantation surgery at Johns Hopkins Hospital..

Design:

* This study will require one visit of approximately 4 to 6 hours.
* Participants will be screened with a full physical examination and medical history, along with a basic hearing test.
* Participants will have a magnetic resonance imaging (MRI) scan of the brain, followed by a MEG scan to record magnetic field changes produced by brain activity.
* During MEG recording, participants will be asked to listen to various sounds and make simple responses (pressing a button, moving your hand or speaking) in response to sounds heard through earphones. The MEG procedure should take between 1 and 2 hours.
* Treatment at NIH is not provided as part of this protocol.

DETAILED DESCRIPTION:
Objective: Auditory processing disorders are common in patients with epilepsy and adversely impact verbal communication. The neural bases of auditory disorders remain poorly understood, impeding development of objective clinical tests. The overall goal of this project is to develop an objective clinical measure of auditory processing using computational modeling of functional brain connectivity. To address this goal, we will use novel functional connectivity methods to analyze magnetoencephalographic (MEG) and intracranial electrocorticographic (ECoG) recordings.

Study Population: We will acquire MEG data from 48 patients with intractable epilepsy prior to their undergoing grid electrode placement for neurosurgery evaluation at Johns Hopkins Hospital. ECoG data will be acquired at JHU under an ongoing study. Approximately half the patients will have auditory processing impairments. We will also acquire MEG from 20 healthy control subjects with no auditory processing impairment.

Design: Three planned studies use a within-subject, repeated measures design. The MEG studies will be conducted before patients have subdural electrodes implanted for intracranial mapping. The MEG studies and connectivity analyses will be performed at NIH. The ECoG studies will take place at Johns Hopkins Hospital. Data will be acquired using the same auditory stimuli and tasks for both the MEG and ECoG parts of the study. The same functional connectivity analyses will be performed on the two data sets.

Outcome measures: The main outcome measures will be (1) functional connectivity patterns in intracranial ECoG data that differentiate epilepsy patients with auditory impairments from those without auditory impairments; and (2) corresponding patterns in MEG data. Secondary outcome measures will consist of relationships between the intracranial ECoG connectivity measures and the MEG connectivity measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal peripheral hearing: pure tone air conduction thresholds less than or equal to 20 dB HL at octave frequencies between 250-8000 Hz for each ear; word recognition scores in quiet greater than or equal to 88% for each ear; normal 226 Hz tympanometry (middle ear peak pressure at 0 plus/minus 100 daPa and peak compensated static compliance of 0.3-1.5 mmho); no history of chronic otitis media, PE tubes, or hearing loss

For those participants with epilepsy - seizure onset age > 10 years

Normal cognitive function (Full-Scale IQ >84)

Absence of any co-morbid neurological disorder

Absence of highly magnetizable metallic implants, including highly magnetizable dental work

A negative urine pregnancy test

For participants with epilepsy scheduled or to-be-scheduled for grid implantation surgery at Johns Hopkins Hospital

EXCLUSION CRITERIA:

Evidence of neurological or psychiatric disorder that would interfere with data interpretation, including cognitive impairment

Presence of a lesion on a previous MRI, except for the following: mesotemporal sclerosis, cortical dysplasia, and dysembryoplastic neuroepithelial tumor.

Presence of highly magnetizable metallic implants, such as pacemakers, aneurysm clips, cochlear implants and shrapnel fragments, including highly magnetizable dental work, or any significant history of exposure to small metallic objects which may have become lodged in the head or neck.

For controls (healthy volunteers) only: history of speech-language disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09-10; Study Completion 2017-04-04

PRIMARY OUTCOMES:
The main outcome measures were to be (1) functional connectivity patterns in intracranial ECoG data that differentiate epilepsy patients with auditory impairments from those without auditory impairments; and (2) corresponding patterns in ... | 12-18 months

SECONDARY OUTCOMES:
Secondary outcome measures were to consist of relationships between the intracranial ECoG connectivity measures and the MEG connectivity measures. | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Horwitz, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Axmacher N, Schmitz DP, Wagner T, Elger CE, Fell J. Interactions between medial temporal lobe, prefrontal cortex, and inferior temporal regions during visual working memory: a combined intracranial EEG and functional magnetic resonance imaging study. J Neurosci. 2008 Jul 16;28(29):7304-12. doi: 10.1523/JNEUROSCI.1778-08.2008. PMID 18632934
- [Background] Babiloni C, Bares M, Vecchio F, Brazdil M, Jurak P, Moretti DV, Ubaldi A, Rossini PM, Rektor I. Synchronization of gamma oscillations increases functional connectivity of human hippocampus and inferior-middle temporal cortex during repetitive visuomotor events. Eur J Neurosci. 2004 Jun;19(11):3088-98. doi: 10.1111/j.0953-816X.2004.03431.x. PMID 15182317
- [Background] Bishop DV, McArthur GM. Individual differences in auditory processing in specific language impairment: a follow-up study using event-related potentials and behavioural thresholds. Cortex. 2005 Jun;41(3):327-41. doi: 10.1016/s0010-9452(08)70270-3. PMID 15871598